CLINICAL TRIAL: NCT05745844
Title: Management of Patients Under Anti-HORMonal Treatment for Prostate Cancer : Evaluation of Neuromuscular ElectroStimulation in Addition to a Physical Activity Program
Brief Title: Evaluation of Neuromuscular ElectroStimulation in Addition to a Physical Activity Program
Acronym: HORMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A00904-39
Record Dates: First submitted 2023-02-14; First posted 2023-02-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, open-label, comparative (two arms), randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroMuscular Electro Stimulation group (Experimental): Patients in the NeuroMuscular Electro Stimulation group will also have neurostimulation sessions using a CE marked medical device, in its destination, according to its instructions for use, therefore without expected clinical risk
  Interventions: Other: activity sessions
- Control Group (Active Comparator): The control group (without NeuroMuscular Electro Stimulation) corresponds to the standard care routinely offered to patients in the investigating centre.
  Interventions: Other: activity sessions

INTERVENTIONS:
Other: activity sessions — 77 activity sessions ; muscle strengthening, testing or unloading

SUMMARY:
The purpose of the study is to measure the muscle strength of the quadriceps 6 months from the start of the intervention, either the maximum load resistance that can be lifted in a single repetition under standardized conditions with the thigh press.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, open, comparative (two arms), randomized, monocentric study, focusing on a therapeutic strategy (muscle strengthening program with or without NeuroMuscular ElectroStimulation).

Patients will be cared for according to a nutritional and sports support program offered routinely in the investigating center, which corresponds to the recommendations for the care of patients with prostate cancer under Androgen Deprivation Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with pharmacological androgen deprivation therapy for prostate cancer for more than 26 weeks;
* Performance index (WHO): 0 or 1;
* Patient able to understand the information related to the study, to read the information leaflet and having consented to participate in the study;
* Patient benefiting from a social security scheme;

Exclusion Criteria:

* Weight ≥ 130 kg;
* Vegetarian food;
* Other associated neoplasia;
* Patient having undergone a bilateral orchiectomy;
* Painful bone metastases, or at risk of fracture;
* Anemia (hemoglobin < 10 g/dL);
* Thrombocytopenia (platelets < 50 G/L);
* Renal impairment (creatinine clearance < 60 mL/min, or albuminuria > 30);
* Patient planning to travel more than 4 weeks continuously in the next 52 weeks;
* Absolute contraindication to physical training (e.g. musculoskeletal, cardiovascular or neurological disorders), according to the doctor specializing in the associated medical condition;
* Contraindication to the use of the neuromuscular electrostimulation device or the impedance meter, in particular infectious disease in the acute phase, fungal infection, dermatitis, unbalanced arrhythmia, epilepsy, wearing an active implantable device (pacemaker, heart artificial, prosthesis incorporating an electromagnetic system), open wound;
* Sports activity already supervised by a third party or at an equal or higher level than the bodybuilding/muscle strengthening work recommended in the study;
* Protected adult patient (under guardianship or curatorship, or under a regime of deprivation of liberty);
* Patient participating in another research, or in a period of exclusion from another research.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle strength | 6 months
  Muscular strength of the quadriceps at 6 months from the start of the intervention, i.e. the maximum resistance / load that can be lifted in a single repetition, under standardized conditions.
  The main analysis is the comparison of quadriceps muscle strength (Maximum Resistance raised in 1 repetition) at 6 months between the groups with neuromuscular electrical stimulation and without neuromuscular electrical stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé Pays de Savoie, Annemasse, France

IPD SHARING:
Plan to Share IPD: No